CLINICAL TRIAL: NCT00826280
Title: A Phase 3b, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Effect of Caffeine Intake on Single Photon Emission Computed Tomography (SPECT) Myocardial Perfusion Imaging (MPI) in Subjects Administered Regadenoson
Brief Title: Caffeine's Effect on Regadenoson Administration With Single Photon Emission Computed Tomography (SPECT) Myocardial Perfusion Imaging (MPI)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 3606-CL-3002
Record Dates: First submitted 2009-01-21; First posted 2009-01-22 (Estimated); Results first posted 2011-10-21 (Estimated); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Coronary Artery Disease (CAD)
Keywords: pharmacologic stress; ischemia; coronary artery disease (CAD)
MeSH Terms: conditions — Coronary Artery Disease; Ischemia | interventions — regadenoson; Technetium; Technetium Tc 99m Sestamibi; technetium tc-99m tetrofosmin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo plus Regadenoson (Placebo Comparator): Two placebo capsules plus 0.4 mg regadenoson per 5mL intravenous (IV) bolus injection
  Interventions: Drug: regadenoson; Radiation: technetium; Drug: placebo
- Caffeine 200 mg plus Regadenoson (Experimental): One 200 mg Caffeine capsule and one placebo capsule plus 0.4 mg regadenoson per 5mL intravenous bolus injection
  Interventions: Drug: regadenoson; Drug: overencapsulated caffeine; Radiation: technetium
- Caffeine 400 mg plus Regadenoson (Experimental): Two 200 mg Caffeine capsules plus 0.4 mg regadenoson per 5mL intravenous bolus injection
  Interventions: Drug: regadenoson; Drug: overencapsulated caffeine; Radiation: technetium

INTERVENTIONS:
Drug: regadenoson — IV
  Other Names: Lexiscan; CVT 3146
Drug: overencapsulated caffeine — oral
  Arms: Caffeine 200 mg plus Regadenoson; Caffeine 400 mg plus Regadenoson
Radiation: technetium — IV
  Other Names: sestamibi; tetrafosmin
Drug: placebo — oral
  Arms: Placebo plus Regadenoson

SUMMARY:
Observe whether the administration of caffeine prior to regadenoson will affect the interpretation of test results in subjects with coronary artery disease (CAD) undergoing SPECT MPI

DETAILED DESCRIPTION:
All subjects will undergo rest and stress scans. Those subjects who qualify by demonstrating at least 1 reversible defect, will undergo a third scan. All stress scans will involve the injection of regadenoson as the pharmacologic stress agent. Prior to the third scan, the subject will be administered blinded capsules of placebo or caffeine.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have undergone a previous diagnostic study [e.g., SPECT, echocardiography, magnetic resonance imaging (MRI), etc.] for a clinical indication demonstrating evidence of reversible defects in ≥ 1 vascular segment, have had other stress testing within the past 3 months, or the subject's history suggests at least a 50% likelihood of CAD

  * If the previous diagnostic study shows only 1 reversible defect and it is in segment 17, another reversible defect will need to be present
* Subject with CAD must have an intermediate/low-risk for immediate intervention
* Subject must ingest caffeinated food or beverages regularly (at least the equivalent of one cup of caffeinated coffee daily)
* Subject must agree to not ingest any caffeine or other foods containing methylxanthine at least 24 hours prior to each study visit
* Subject must agree to abstain from eating solid food or drinking liquids other than water for at least 30 minutes prior to each study visit and 30 minutes following each study visit

Exclusion Criteria:

* Subject with documented myocardial infarction (MI) ≤ 30 days prior to enrollment
* Subject with history of percutaneous coronary intervention (PCI) ≤ 4 weeks prior to enrollment
* Subject with history of coronary artery bypass graft (CABG) ≤ 8 weeks prior to enrollment
* Subject has prior history of heart transplantation
* Subject has unstable angina, known severe left main coronary artery stenosis, severe heart failure, uncontrolled arrhythmias, symptomatic hypotension or severe hypertension (systolic blood pressure < 90 or > 180 mmHg, respectively), or > 1st degree atrioventricular block in the absence of a functioning pacemaker
* Subject requires emergent cardiac medical intervention or catheterization
* Subject has a history of smoking, regardless of frequency, tobacco type or method of intake, or using any smoking cessation products, including but not limited to the nicotine patch or nicotine gum, within 3 months prior to first dose of regadenoson
* Subject is currently undergoing treatment with theophylline, or theophylline containing medications within 7 days prior to randomization (Day 3)
* Subject has a history of known or suspected bronchoconstrictive or bronchospastic lung disease [e.g., asthma, wheezing, chronic obstructive pulmonary disease (COPD), etc.]
* Subject has a history of diabetes associated with gastric disorders and/or emptying
* Subject has end stage renal disease (ESRD) with a GFR< 15mL/min or currently undergoing dialysis for ESRD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 347 (Actual)
Dates: Start 2009-03-24 (Actual); Primary Completion 2010-07-15 (Actual); Study Completion 2010-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma Global Development
Locations (25):
- United States (25):
  - Birmingham, Alabama
  - Huntsville, Alabama
  - La Mesa, California
  - Mission Viejo, California
  - Roseville, California
  - Sacramento, California
  - Santa Rosa, California
  - Hartford, Connecticut
  - Newark, Delaware
  - Jacksonville, Florida
  - Miami, Florida
  - Tamarac, Florida
  - Aurora, Illinois
  - Overland Park, Kansas
  - Auburn, Maine
  - Pittsfield, Massachusetts
  - Detroit, Michigan
  - Ypsilanti, Michigan
  - Kansas City, Missouri
  - Albany, New York
  - Rochester, New York
  - Columbus, Ohio
  - Philadelphia, Pennsylvania
  - Wyomissing, Pennsylvania
  - Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Tejani FH, Thompson RC, Iskandrian AE, McNutt BE, Franks B. Effect of caffeine on SPECT myocardial perfusion imaging during regadenoson pharmacologic stress: rationale and design of a prospective, randomized, multicenter study. J Nucl Cardiol. 2011 Feb;18(1):73-81. doi: 10.1007/s12350-010-9311-6. Epub 2010 Nov 17. PMID 21082298
- See also: Link to results on Astellas Clinical Study Results website — https://www.astellasclinicalstudyresults.com/study.aspx?ID=49

RESULTS

PARTICIPANT FLOW:
Groups:
- Caffeine 400 mg Plus Regadenoson: Two 200 mg Caffeine capsule plus 0.4 mg regadenoson per 5mL intravenous bolus injection
Period: Overall Study
Arm/Group | Placebo Plus Regadenoson | Caffeine 200 mg Plus Regadenoson | Caffeine 400 mg Plus Regadenoson
Started | 114 | 116 | 117
Safety Analysis Set | 113 (Safety Analysis Set (SAF) was all randomized subjects who received at least one dose of regadenoson) | 116 (SAF was all randomized subjects who received at least one dose of regadenoson) | 116 (SAF was all randomized subjects who received at least one dose of regadenoson)
Completed Treatment | 66 (Subjects who completed treatment but had ≥ 1 non-interpretable scan were not included in FAS) | 71 (Subjects who completed treatment but had ≥ 1 non-interpretable scan were not included in FAS) | 72 (Subjects who completed treatment but had ≥ 1 non-interpretable scan were not included in FAS)
Completed | 66 (Ending Population equals FAS, all randomized subjects with interpretable MPI scans) | 70 (Ending Population equals FAS, all randomized subjects with interpretable MPI scans) | 71 (Ending Population equals FAS, all randomized subjects with interpretable MPI scans)
Not Completed | 48 | 46 | 46
Not completed — Randomized but drug not received | 1 | 0 | 1
Not completed — Adverse Event | 1 | 3 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Sponsor discontinued subject or study | 1 | 0 | 0
Not completed — Reversible ischemic defect not present | 43 | 40 | 44
Not completed — Interpretation Failure | 1 | 0 | 0
Not completed — Machine Failure | 1 | 1 | 0
Not completed — One or more non-interpretable scan | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Plus Regadenoson | Caffeine 200 mg Plus Regadenoson | Caffeine 400 mg Plus Regadenoson | Total
Number analyzed (Participants) | 66 | 70 | 71 | 207
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.0 (9.99) | 65.7 (11.11) | 69.4 (8.23) | 67.7 (9.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 20 | 43
  Male | 55 | 58 | 51 | 164
Race/Ethnicity, Customized [Number; unit: participants]
  White | 61 | 63 | 68 | 192
  Black or African American | 5 | 5 | 3 | 13
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Number of Reversible Defects
Description: Each segment of the 17-Segment Model was assessed for radiotracer uptake on a scale of 0 (normal uptake) to 4 (absent uptake). Segments were counted as having a reversible defect if the stress score was greater than the rest score and the stress score was ≥ 2. Change was calculated as the number of reversible defects using regadenoson with caffeine/placebo (Day 5) minus the number of reversible defects using regadenoson alone (Day 3).
Time Frame: Day 3 and Day 5
Population: The number of participants analyzed represents Full Analysis Set (FAS), which included all randomized subjects with interpretable Myocardial Perfusion Imaging (MPI) scans. The number of participants per arm is consistent for all categories of the data table.
Measure: Mean (Standard Deviation); unit: Reversible Defects
Arm/Group | Placebo Plus Regadenoson | Caffeine 200 mg Plus Regadenoson | Caffeine 400 mg Plus Regadenoson
Number analyzed (Participants) | 66 | 70 | 71
Reversible Defects
  Baseline Stress Scan (Day 3) | 0.67 (1.377) | 1.01 (1.452) | 1.00 (1.595)
  Double-Blind Stress Scan (Day 5) | 0.80 (1.511) | 0.40 (0.907) | 0.38 (0.962)
  DoubleBlind - Baseline (Day 5 - Day 3) | 0.12 (0.981) | -0.61 (1.097) | -0.62 (1.367)
Statistical Analysis 1: Comparison: Placebo Plus Regadenoson vs Caffeine 200 mg Plus Regadenoson vs Caffeine 400 mg Plus Regadenoson; P-Value applies to 'Double-Blind - Baseline (Day 5 - Day 3)'; Test type: Superiority or Other; p < 0.001, ANCOVA — P-Value is from the primary analysis using ANCOVA
Statistical Analysis 2: Comparison: Placebo Plus Regadenoson vs Caffeine 200 mg Plus Regadenoson; P-Value applies to 'Double-Blind - Baseline (Day 5 - Day 3)'; Test type: Superiority or Other; p < 0.001, ANCOVA — The unadjusted P-Values for pairwise differences should be used for interpretation only if the treatment effect's P-Value ≤ 0.05
Statistical Analysis 3: Comparison: Placebo Plus Regadenoson vs Caffeine 400 mg Plus Regadenoson; P-Value applies to 'Double-Blind - Baseline (Day 5 - Day 3)'; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: Caffeine 200 mg Plus Regadenoson vs Caffeine 400 mg Plus Regadenoson; P-Value applies to 'Double-Blind - Baseline (Day 5 - Day 3)'; Test type: Superiority or Other; p = 0.9328, ANCOVA — [p-value comment as in outcome 1, analysis 2]

2. Secondary Outcome: Change in Summed Difference Score (SDS) Across All 17 Segments
Description: The Summed Difference Score was calculated as the difference in the Summed Stress Score across the 17 segments (scan run under stress condition) minus the Summed Rest Score across the 17 segments (scan run under rest conditions). Change in SDS was calculated as the SDS for regadenoson with caffeine/placebo stress scan (Day 5) minus the SDS for regadenoson only stress scan (Day 3). The full range of the SDS is -68 to 68, where 0 represents no change between Summed Stress Score and Summed Rest Score. A higher positive score indicates more severe coronary artery disease (CAD).
Time Frame: Day 3 and Day 5
Population: The number of participants analyzed represents Full Analysis Set (FAS), which included all randomized subjects with interpretable MPI scans. The number of participants per arm is consistent for all categories of the data table.
Measure: Mean (Standard Deviation); unit: Sum Difference Score
Arm/Group | Placebo Plus Regadenoson | Caffeine 200 mg Plus Regadenoson | Caffeine 400 mg Plus Regadenoson
Number analyzed (Participants) | 66 | 70 | 71
Sum Difference Score
  Baseline Stress Scan (Day 3) | 2.24 (3.013) | 2.45 (2.909) | 2.53 (3.086)
  Double-Blind Stress Scan (Day 5) | 2.36 (3.247) | 1.42 (2.091) | 1.27 (2.003)
  DoubleBlind - Baseline (Day 5 - Day 3) | 0.11 (2.871) | -1.03 (2.071) | -1.25 (2.664)
Statistical Analysis 1: Comparison: Placebo Plus Regadenoson vs Caffeine 200 mg Plus Regadenoson vs Caffeine 400 mg Plus Regadenoson; P-Value applies to 'Double-Blind - Baseline (Day 5 - Day 3)'; Test type: Superiority or Other; p = 0.0011, ANCOVA — P-Value is from the primary analysis using ANCOVA
Statistical Analysis 2: Comparison: Placebo Plus Regadenoson vs Caffeine 200 mg Plus Regadenoson; P-Value applies to 'Double-Blind - Baseline (Day 5 - Day 3)'; Test type: Superiority or Other; p = 0.0034, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo Plus Regadenoson vs Caffeine 400 mg Plus Regadenoson; P-Value applies to 'Double-Blind - Baseline (Day 5 - Day 3)'; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: Caffeine 200 mg Plus Regadenoson vs Caffeine 400 mg Plus Regadenoson; P-Value applies to 'Double-Blind - Baseline (Day 5 - Day 3)'; Test type: Superiority or Other; p = 0.5902, ANCOVA — [p-value comment as in outcome 1, analysis 2]

3. Secondary Outcome: Change in Number of Reversible Defects Assessed by Computerized Quantitation
Description: as for outcome 1
Time Frame: Day 3 and Day 5
Population: The number of participants analyzed per arm represents Full Analysis Set (FAS), all randomized subjects with interpretable MPI scans. The number of participants included in the calculation for each visit is noted in the category titles, as "N".
Measure: Mean (Standard Deviation); unit: Reversible Defects
Arm/Group | Placebo Plus Regadenoson | Caffeine 200 mg Plus Regadenoson | Caffeine 400 mg Plus Regadenoson
Number analyzed (Participants) | 66 | 70 | 71
Reversible Defects
  Baseline Stress Scan (Day 3) [N=64; 69; 70] | 1.47 (1.927) | 2.00 (2.364) | 2.19 (2.122)
  Double-Blind Stress Scan (Day 5) [N=66; 70; 71] | 1.74 (2.355) | 1.46 (1.954) | 1.42 (1.794)
  DoubleBlind - Baseline (Day 5-Day 3)[N=64; 69; 70] | 0.31 (1.622) | -0.59 (1.743) | -0.81 (1.812)
Statistical Analysis 1: Comparison: Placebo Plus Regadenoson vs Caffeine 200 mg Plus Regadenoson vs Caffeine 400 mg Plus Regadenoson; P-Value applies to 'Double-Blind - Baseline (Day 5 - Day 3)'; Test type: Superiority or Other; p = 0.0037, ANCOVA — P-Value is from the primary analysis using ANCOVA
Statistical Analysis 2: Comparison: Placebo Plus Regadenoson vs Caffeine 200 mg Plus Regadenoson; P-Value applies to 'Double-Blind - Baseline (Day 5 - Day 3)'; Test type: Superiority or Other; p = 0.0089, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo Plus Regadenoson vs Caffeine 400 mg Plus Regadenoson; P-Value applies to 'Double-Blind - Baseline (Day 5 - Day 3)'; Test type: Superiority or Other; p = 0.0016, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: Caffeine 200 mg Plus Regadenoson vs Caffeine 400 mg Plus Regadenoson; P-Value applies to 'Double-Blind - Baseline (Day 5 - Day 3)'; Test type: Superiority or Other; p = 0.5654, ANCOVA — [p-value comment as in outcome 1, analysis 2]

4. Secondary Outcome: Change in Summed Difference Score Across All 17 Segments Assessed by Computerized Quantitation
Description: as for outcome 2
Time Frame: Day 3 and Day 5
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Summed Difference Score
Arm/Group | Placebo Plus Regadenoson | Caffeine 200 mg Plus Regadenoson | Caffeine 400 mg Plus Regadenoson
Number analyzed (Participants) | 66 | 70 | 71
Summed Difference Score
  Baseline Stress Scan (Day 3) [N=64; 69; 70] | 3.34 (4.383) | 4.46 (4.604) | 4.29 (4.314)
  Double-Blind Stress Scan (Day 5) [N=66; 70; 71] | 4.41 (4.874) | 3.10 (4.737) | 2.46 (3.601)
  DoubleBlind - Baseline (Day 5-Day 3)[N=64; 69; 70] | 1.02 (3.364) | -1.45 (3.890) | -1.84 (3.658)
Statistical Analysis 1: Comparison: Placebo Plus Regadenoson vs Caffeine 200 mg Plus Regadenoson vs Caffeine 400 mg Plus Regadenoson; P-Value applies to 'Double-Blind - Baseline (Day 5 - Day 3)'; Test type: Superiority or Other; p < 0.001, ANCOVA — P-Value is from the primary analysis using ANCOVA
Statistical Analysis 2: Comparison: Placebo Plus Regadenoson vs Caffeine 200 mg Plus Regadenoson; P-Value applies to 'Double-Blind - Baseline (Day 5 - Day 3)'; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo Plus Regadenoson vs Caffeine 400 mg Plus Regadenoson; P-Value applies to 'Double-Blind - Baseline (Day 5 - Day 3)'; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: Caffeine 200 mg Plus Regadenoson vs Caffeine 400 mg Plus Regadenoson; P-Value applies to 'Double-Blind - Baseline (Day 5 - Day 3)'; Test type: Superiority or Other; p = .4246, ANCOVA — [p-value comment as in outcome 1, analysis 2]

5. Secondary Outcome: Change From Baseline in Heart Rate
Description: Baseline is the last non-missing measurement on or before first dose of regadenoson Change is calculated as the time point minus baseline.
Time Frame: Baseline, Day 5 (-3 min), Day 5 (+3 min), Day 5 (+15 min)
Population: The number of participants analyzed per arm represents Safety Analysis Set (SAF) all randomized patients who received at least one dose of regadenoson. The number of participants included in the calculation for each visit is noted in the category titles, as "N".
Measure: Median (Full Range); unit: Beats per minute
Arm/Group | Placebo Plus Regadenoson | Caffeine 200 mg Plus Regadenoson | Caffeine 400 mg Plus Regadenoson
Number analyzed (Participants) | 113 | 116 | 116
Beats per minute
  Baseline [N=113; 116; 116] | 66.0 [46 to 96] | 62.0 [45 to 92] | 64.0 [47 to 97]
  Change at Day 5 (- 3 min) [N=67; 70; 71] | -2.0 [-23 to 51] | -1.0 [-29 to 75] | -2.0 [-22 to 11]
  Change at Day 5 (+3 min) [N=67; 70; 72] | 9.0 [-20 to 38] | 5.0 [-23 to 58] | 0.0 [-16 to 22]
  Change at Day 5 (+15 min) [N=66; 72; 72] | 4.0 [-19 to 31] | 1.0 [-21 to 63] | -1.0 [-20 to 25]

6. Secondary Outcome: Change From Baseline in Systolic Blood Pressure
Description: Baseline is the last non-missing measurement on or before first dose of regadenoson. Change is calculated as the time point minus baseline.
Time Frame: Baseline, Day 5 (-3 min), Day 5 (+3 min), Day 5 (+15 min)
Population: as for outcome 5
Measure: Median (Full Range); unit: mmHg
Arm/Group | Placebo Plus Regadenoson | Caffeine 200 mg Plus Regadenoson | Caffeine 400 mg Plus Regadenoson
Number analyzed (Participants) | 113 | 116 | 116
mmHg
  Baseline [N=113; 116; 116] | 135.0 [95 to 184] | 131.0 [88 to 180] | 135.0 [100 to 179]
  Change at Day 5 (- 3 min) [N=67;70;71] | 0.0 [-26 to 46] | 12.0 [-35 to 58] | 11.0 [-20 to 46]
  Change at Day 5 (+3 min) [N=67; 70; 72] | 0.0 [-37 to 36] | 8.0 [-42 to 52] | 7.5 [-25 to 44]
  Change at Day 5 (+15 min) [N=66; 72; 72] | -2.0 [-37 to 37] | 8.0 [-30 to 68] | 5.0 [-26 to 46]

7. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure
Description: as for outcome 6
Time Frame: Baseline, Day 5 (-3 min), Day 5 (+3 min), Day 5 (+15 min)
Population: as for outcome 5
Measure: Median (Full Range); unit: mmHg
Arm/Group | Placebo Plus Regadenoson | Caffeine 200 mg Plus Regadenoson | Caffeine 400 mg Plus Regadenoson
Number analyzed (Participants) | 113 | 116 | 116
mmHg
  Baseline [N= 113; 116;116] | 78.0 [45 to 100] | 74.0 [48 to 102] | 73.0 [51 to 106]
  Change at Day 5 (- 3 min) [N=67; 70; 71] | 0.0 [-22 to 14] | 4.0 [-19 to 20] | 6.0 [-12 to 47]
  Change at Day 5 (+ 3 min) [N=67; 70; 72] | -1.0 [-19 to 23] | 4.0 [-20 to 30] | 3.0 [-22 to 28]
  Change at Day 5 (+15 min) [N=66; 72; 72] | -2.0 [-26 to 18] | 3.0 [-18 to 23] | 4.0 [-16 to 41]

ADVERSE EVENTS:
Time Frame: Beginning of Day 3 through the Day 6 visit. All Serious Adverse Events occurring until 30 days after dosing were to be reported.
Description: Any untoward medical occurrence that occurred at the beginning of day 3 (Baseline Stress Scan) through the day 6 visit (considered "treatment- emergent") was recorded as an Adverse Event. Within a system organ class subjects may have reported more than one type of Adverse Event.
Arm/Group | Placebo Plus Regadenoson | Caffeine 200 mg Plus Regadenoson | Caffeine 400 mg Plus Regadenoson
Serious Adverse Events (participants affected / at risk) | 1/113 | 2/116 | 2/116
Other Adverse Events (participants affected / at risk) | 82/113 | 89/116 | 80/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Plus Regadenoson (N=113) | Caffeine 200 mg Plus Regadenoson (N=116) | Caffeine 400 mg Plus Regadenoson (N=116)
Angina pectoris (Cardiac disorders) | 1 | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 1
Myocardial infraction (Cardiac disorders) | 0 | 1 | 0
Acute myocardial infraction (Cardiac disorders) | 0 | 0 | 1
Renal failure acute (Cardiac disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Plus Regadenoson (N=113) | Caffeine 200 mg Plus Regadenoson (N=116) | Caffeine 400 mg Plus Regadenoson (N=116)
Abdominal discomfort (Gastrointestinal disorders) | 6 | 3 | 5
Abdominal pain upper (Gastrointestinal disorders) | 6 | 4 | 5
Nausea (Gastrointestinal disorders) | 13 | 16 | 10
Stomach discomfort (Gastrointestinal disorders) | 7 | 4 | 4
Chest discomfort (General disorders) | 22 | 25 | 19
Chest pain (General disorders) | 8 | 1 | 2
Feeling hot (Gastrointestinal disorders) | 3 | 5 | 6
Dizziness (Nervous system disorders) | 22 | 25 | 18
Dysgeusia (Nervous system disorders) | 4 | 11 | 5
Headache (Nervous system disorders) | 36 | 37 | 38
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 43 | 47 | 34
Flushing (Vascular disorders) | 27 | 29 | 27

LIMITATIONS AND CAVEATS:
Company makes no warranties or representations of any kind as to the posting, expressed or implied, including warranties of merchantability and fitness for a particular purpose, and shall not be liable for any damages.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript at least 30 days prior to publication to ensure that no confidential information of Sponsor is included in the document. Sponsor may delay the publication for an additional 60 days to seek patent protection.